CLINICAL TRIAL: NCT02427529
Title: Muscle-Sparing Effect Of Human Chorionic Gonadotropin (hCG) During a Very Low Calorie Diet (VLCD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Emma's Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 053111
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: HCG
Keywords: hcg
MeSH Terms: conditions — Hypertrichosis congenital generalized X-linked | interventions — Chorionic Gonadotropin; Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCG Group (Experimental): This group received daily subcutaneous injections of Human Chorionic Gonadotropin while eating a very low calorie diet of 500 calories per day.
  Interventions: Drug: Human Chorionic Gonadotropin; Other: Low calorie diet
- Saline/Placebo (Placebo Comparator): This group received daily subcutaneous injections of saline while eating a very low calorie diet of 500 calories per day.
  Interventions: Drug: Placebo; Other: Low calorie diet

INTERVENTIONS:
Drug: Human Chorionic Gonadotropin — The addition of hormone to a daily low calorie diet to potentially aid in selective fat loss, or muscle-sparing.
  Other Names: Pregnyl, Novarel
  Arms: HCG Group
Drug: Placebo
  Arms: Saline/Placebo
Other: Low calorie diet

SUMMARY:
Subjects are female patients, randomized to HCG group or placebo group, during a prospective trial, in order to determine the significance, if any, of HCG on maintaining muscle mass during a very low calorie diet in order to demonstrate the potential significance of HCG administration on preserving lean body mass while losing weight.

DETAILED DESCRIPTION:
Four-week clinical trials were conducted on 59 females between the ages of 20 and 55, over an 18 month period. Exclusion criteria included thyroid conditions or prior significant medical history. Patients were randomized to receive daily subcutaneous injections of either hCG (200-300IU) or saline (placebo). All were placed on a VLCD resembling a protein-sparing modified fast. The caloric intake was between 500 and 600 calories, with 50% protein and 50% complex carbohydrates consisting mostly of fruits and vegetables. Measured parameters: weight, body composition via bio-impedance, blood pressure, and blood labs. A subset also underwent weekly electrocardiograms (EKG).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than 30,
* Female,
* good health

Exclusion Criteria:

* complex medical history,
* thyroid disease,
* BMI less than 30,
* psychological instability or history of eating disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight loss achieved during a trial of HCG vs. Placebo and a very low calorie diet. | 30 days
  Comparison of weight loss between the experimental and control group

SECONDARY OUTCOMES:
Muscle loss comparison between HCG and placebo group during a very low calorie diet. | 30 days
  Lean body mass and muscle mass readings used to compare between experimental and control group.

OTHER OUTCOMES:
Fat loss comparison between HCG and placebo groups during a very low calorie diet. | 30 days
  Fat mass readings used to compare between experimental and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Emma's Corporation, Colts Neck, New Jersey, United States